CLINICAL TRIAL: NCT05919628
Title: Psychological Ressources as a Protective Factor for Anxiety-depression, Well-being and Therapeutical Observance in Parkinson's Disease.
Brief Title: Psychological Ressources, Anxiodepressive Symptoms, Well-being and Therapeutical Observance in Parkinson's Disease
Acronym: ResPsyPark
Status: Completed | Type: Observational
Sponsor: Central Hospital, Nancy, France (Other)
Responsible Party: Principal Investigator, Mme Mylène MEYER, Psychologist, PhD, Central Hospital, Nancy, France
Other Study IDs: 2023PI077
Record Dates: First submitted 2023-05-19; First posted 2023-06-26 (Actual); Last update posted 2023-09-06 (Actual); Status verified 2023-09

CONDITIONS: Parkinson's Disease
Keywords: psychological ressources; well-being; depression; anxiety; therapeutical observance; parkinson's disease
MeSH Terms: conditions — Parkinson Disease; Depression; Anxiety Disorders

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: ResPsyPark group — Evaluation of the parkinson's disease patient's score over different psychological questionnaires and a therapeutical observance questionnaire

SUMMARY:
Anxiodepressive symptoms are frequently observed in Parkinson's disease patients. These non motor psychiatric charateristics of the disease negatively impairs quality of life, and may impair well-being or therapeutical observance.

The objective of this study is to determine if psychological ressources are associated to anxiodepressive symptoms, to parkinson well-being and therapeutical observance. It will be interesting to determine if the presence of some - or multiple- psychological ressources could prevent patients from anxiety, depression, impaired well-being and impaired observance.

This study will analyse retrospectively psychological scalescompleted by 30 parkinson's disease patients through previous psychological interviews. The scales investigate anxiety, depression, well-being, psychological ressources, and therapeutical observance.

The results will highlight the importance of working on psychological ressources with Parkinson's disease patients through psychotherapy, in order to improve their well-being, positive emotions and maybe contribute to better therapeutical observance.

DETAILED DESCRIPTION:
The scales used are :

* The SPANE
* The PAS
* The LOT-R
* The SCS
* The brief BDI
* The SSAM
* The HAD
* The MAAS
* An observance scale

ELIGIBILITY:
Inclusion Criteria:

* Patients with diagnosis of Parkinson's disease

Exclusion Criteria:

* Patients with any other parkinsonian syndrome

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Parkinson's disease patients at any stage of the disease.
Sampling Method: Non-Probability Sample
Enrollment: 25 (Actual)
Dates: Start 2023-06-15 (Actual); Primary Completion 2023-06-15 (Actual); Study Completion 2023-06-30 (Actual)

PRIMARY OUTCOMES:
Study of the links between psychological ressources and anxiodepressive symptoms | At baseline
  Correlation and regression analysis between scores at the scales evaluating anxiety (PAS, HAD) and depression (BDI, HAD), and scores at the scales evaluating psychological ressources (LOT-R, SCS, SSAm, MAAS).

SECONDARY OUTCOMES:
Study of the links between therapeutical observance and anxiodepressive symptoms | At baseline
  Correlation and regression analysis between scores at the scales evaluating anxiety (PAS, HAD) and depression (BDI, HAD), and score at the scale evaluating therapeutical observance (%).

CONTACTS AND LOCATIONS:
Locations (1):
- CHU de Nancy, Nancy, France

IPD SHARING:
Plan to Share IPD: Undecided